CLINICAL TRIAL: NCT04956744
Title: A Phase 1, Dose-Escalating, Open-label Study to Evaluate the Safety, Tolerability, and Exploratory Efficacy of Single Dose of IV IMS001 in Subjects With Multiple Sclerosis and Treatment Failure to Prior Disease Modifying Treatments (DMTs)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Exploratory Efficacy of IMS001 in Subjects With Multiple Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImStem Biotechnology (Industry)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMS001-01
Record Dates: First submitted 2021-06-22; First posted 2021-07-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Low dose of cells/kg of intravenous (IV) IMS001 as a single dose infusion on Day 1.
  Interventions: Biological: IMS001
- High Dose (Experimental): High dose of cells/kg of intravenous (IV) IMS001 as a single dose infusion on Day 1.
  Interventions: Biological: IMS001
- Optional Dose (Experimental): High dose of cells/kg of intravenous (IV) IMS001 as a single dose infusion on Day 1 and at Month 6.
  Interventions: Biological: IMS001

INTERVENTIONS:
Biological: IMS001 — IMS001 is a human embryonic cell derived (hESC) mesenchymal stem cell (MSC).

SUMMARY:
This is a Phase 1 study of IMS001, given as a single dose to subjects with Multiple Sclerosis who experience inadequate response and/or intolerability to disease modifying treatments. IMS001 is a human embryonic cell derived (hESC) mesenchymal stem cell (MSC). MSCs have the potential to modulate disease course.

ELIGIBILITY:
Inclusion Criteria:

* Provides signed and dated informed consent in accordance with local regulations.
* 18 to 65 years of age.
* Diagnosis of MS.
* Has had an inadequate response DMTs.
* EDSS within protocol parameters.
* Able and willing to undergo MRIs.
* Must be clinically stable for 1 month prior to Day 1.

Exclusion Criteria:

* Has a known or suspected hypersensitivity to human serum albumin, diphenhydramine, acetaminophen, methylprednisolone, or any of the components of IMS001.
* Has history of excluded medications, per protocol, prior to Day 1.
* Has a history of neoplastic disease except for basal cell carcinoma, non-metastatic squamous cell carcinoma of the skin that has been excised with clean margins, or adequately treated in-situ carcinoma of the cervix.
* Prior history of any other autoimmune disease, myelodysplasia, or hematologic disease.
* Prior treatment with any allogeneic cell therapy or tissue transplant.
* Prior history of smoking equivalent to ˃20 cumulative pack years of cigarettes.
* Recent clinically significant infection during the Screening Phase.
* Has any medical or psychiatric condition that would impact outcome or participation in the study.
* Has clinically significant abnormal findings on the electrocardiogram (ECG) during the Screening Phase.
* Has known or documented human immunodeficiency virus (HIV) infection or active Hepatitis B, or C.
* Has an elevated liver function test abnormality during the Screening Phase.
* Has abnormalities of blood count during the Screening Phase.
* Has laboratory abnormalities of renal function during the Screening Phase.
* Has other clinically significant laboratory abnormalities during Screening Phase.
* Body weight ≥120 kg.
* Women pregnant, breast feeding, or planning to become pregnant during the study.
* Is unavailable for the duration of the trial, is likely to be noncompliant with the protocol, or is generally felt to be unsuitable by the principal investigator.
* Current or recent participation in any other clinical or device trials within 3 months prior to Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Day 1 to Month 60
  Frequency of treatment-emergent adverse events (TEAEs).
Safety and tolerability | Day 1 to Month 60
  Clinically significant laboratory abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, MD, Study Director — ImStem Biotechnology
Locations (3):
- United States (3):
  - Shepherd Center, Atlanta, Georgia
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Rocky Mountain MS Clinic, Salt Lake City, Utah

REFERENCES:
- See also: Imstem Biotechnology — http://www.imstem.com/